CLINICAL TRIAL: NCT00450385
Title: Phase II Study to Establish Gene Expression Models Predicting Survival of Diffuse Large B-Cell Lymphoma Patients Treated With R-CHOP
Brief Title: Genes in Predicting Outcome of Patients With DLBCL Treated With Rituximab and Combination Chemotherapy (R-CHOP)
Acronym: R-CHOP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator Decision due to insufficient accrual.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Izidore Lossos, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20061138; SCCC-2006069 (Other: University of Miami Sylvester Comprehensive Cancer Center); WIRB-20070073 (Other: Western Institutional Review Board)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-05

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R-CHOP (Experimental): Patients will receive R-CHOP for 6 to 8 cycles:
  * Rituximab 375 mg/m2 on day 1
  * Cyclophosphamide 750 mg/m2 IV on day 1
  * Doxorubicin 50 mg/m2 on day 1
  * Vincristine 1.4 mg/m2 (maximum = 2 mg) IV on day 1
  * Prednisone 100 mg orally days 1-5, repeated every 21 days.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: Vincristine

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m2 on day 1 for 6 to 8 cycles
  Other Names: Rituxan
Drug: Cyclophosphamide — Cyclophosphamide 750 mg/m2 IV on day 1 for 6 to 8 cycles
  Other Names: Cytoxan
Drug: Doxorubicin — Doxorubicin 50 mg/m2 on day 1 for 6 to 8 cycles
  Other Names: Adriamycin
Drug: Prednisone — Prednisone 40 mg/m2 orally days 1-5, repeated every 21 days for 6 to 8 cycles.
  Other Names: Deltasone
Drug: Vincristine — Vincristine 1.4 mg/m2 (maximum = 2 mg) IV on day 1 for 6 to 8 cycles
  Other Names: Oncovin

SUMMARY:
The investigators hypothesize that survival of newly diagnosed DLBCL (diffuse large B-cell lymphoma) patients treated with R-CHOP can be predicted by RNA or protein gene expression or by presence of biomarkers associated with the anti-tumor effects of Rituximab.

DETAILED DESCRIPTION:
In this phase II multi-institutional trial, the investigators will identify genes associated with either good or bad outcome in DLBCL patients treated with R-CHOP, will construct a robust predictive models based on RNA extracted from or paraffin specimens as well on immunohistochemistry and will examine the predictive power of new biomarkers associated with the anti-tumor effects of rituximab. The acquisition of fixed tissue as a component of this uniformly treated prospective study will also afford future studies with this informative dataset.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of diffuse large B-cell lymphoma, CD20-positive, according to the World Health Organization Classification, stages II-IV or limited stage I disease that is bulky (more than 10 cm) or with International Prognostic Index (IPI) score > 1.
* 2. Patients must not have had prior chemotherapy, radiotherapy or immunotherapy. A short course (< 2 weeks) of corticosteroids is allowed.
* 3. Adequate paraffin-embedded tumor specimen must be available for gene expression analysis and immunohistochemistry prior to initiation of therapy. (If the specimen is deemed inadequate, the subject can be retroactively screen failed, as this does not change the treatment regimen).
* 4. Baseline measurements and evaluation must be obtained within 4 weeks before first treatment.
* 5. Age >18 years.
* 6. Eastern Cooperative Oncology Group (ECOG) performance status 0-3.
* 7. Adequate organ function:

  * White Blood Cells count (WBC) >2500/µL
  * Absolute Neutrophil Count (ANC) > 1000/µL (unless due to disease in marrow)
  * platelet count >100,000/µL (unless due to disease in marrow)
  * creatinine < 2.0 mg/dL,
  * bilirubin < 1.5 mg/dL (may be 1.5-3.0 mg/dl if due to liver involvement by lymphoma)
  * Serum Glutamic Oxaloacetic Transaminase (SGOT)/ Serum Glutamic Pyruvic Transaminase (SGPT) <3 x upper limit of normal.
* 8. Female patients must not be pregnant or breast feeding.
* 9. Women of childbearing potential and men must be strongly advised to use an accepted and effective method of contraception.
* 10. Patients must have left ventricular ejection fraction of >45%.
* 11. Provision of written informed consent.

Exclusion Criteria:

* 1. Patients with a second malignancy other than basal cell carcinoma of the skin or in situ carcinoma of the cervix unless the tumor was treated with curative intent at least two years previously; and; the patient continue to be free of evidence of recurrence.
* 2. Patients with HIV infection as these patients are managed on dedicated protocols.
* 3. Patients with active central nervous system (CNS) lymphoma.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-04-24 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Izidore S. Lossos, MD, Study Chair — University of Miami
Locations (5):
- United States (5):
  - Stanford University, Stanford, California
  - University of Miami, Miami, Florida
  - University of Rochester Medical Center - Wilmot Cancer Institute, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 patients were consented, however, only 57 of these patients were found to be eligible for enrollment per the protocol.
Period: Overall Study
Arm/Group | R-CHOP
Started | 57
Completed | 44
Not Completed | 13
Not completed — Death | 3
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Arm/Group | R-CHOP
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Determination of a List of Genes and Construction of Survival Prediction Models That Will Predict Overall Survival at 30 Months in DLBCL Patients Receiving R-CHOP Therapy.
Description: The investigators aim to determine a list of genes and construct survival prediction model(s) that will predict the overall survival at 30 months in DLBCL patients prospectively treated with R-CHOP chemotherapy. Overall survival time will be calculated from the date of the diagnosis until death or last follow-up examination.
Time Frame: 30 months
Population: The study required a minimum of 90 participants for gene expression analyses from which survival prediction model(s) could be derived. Due to actual participant accrual (57) being far below the minimum number of participants required, no data were collected on gene expression, and no survival prediction models were constructed.
Arm/Group | R-CHOP
Number analyzed (Participants) | 0

2. Primary Outcome: Usefulness of Biomarkers Associated With Anti-Tumor Effects of Rituximab in Predicting Overall Survival in DLBCL Patients Receiving R-CHOP Therapy
Description: The investigators aim to determine the usefulness of biomarkers associated with the antitumor effects of rituximab (e.g. immunoglobulin GFc receptor genotypes, CD20 protein expression and gene expression profiles) to predict overall survival of DLBCL patients treated with R-CHOP therapy and followed for at least 24 months or until death.
Time Frame: 24 Months
Population: The study required a minimum of 90 participants for associated biomarker analyses. Due to actual participant accrual (57) being far below the minimum number of participants required, no biomarker data were collected.
Arm/Group | R-CHOP
Number analyzed (Participants) | 0

3. Primary Outcome: Comparison of the Ability of Constructed Survival Models to Predict Overall Survival in DLBCL Patients Receiving R-CHOP Therapy
Description: The investigators will compare the ability of constructed survival models to predict survival in DLBCL patients receiving R-CHOP therapy
Time Frame: 2 Years
Population: The comparison could not be made because the study required a minimum of 90 participants for initial gene expression analyses from which survival prediction model(s) would be derived. Due to actual participant accrual (57) being far below the minimum number of participants required, no gene expression or survival prediction data were collected.
Arm/Group | R-CHOP
Number analyzed (Participants) | 0

4. Secondary Outcome: Determination of the Ability of Models and/or Biomarkers Associated With Anti-Tumor Effects of Rituximab to Predict 24-month Time to Treatment Failure in DLBCL Patients Receiving R-CHOP Therapy
Description: The investigators aim to determine the ability of the models and/or biomarkers associated with the anti-tumor effects of rituximab to predict 24-month time to treatment failure, defined as disease progression, death or initiation of new treatment.
Time Frame: 24 Months
Population: The determination could not be made because the study required a minimum of 90 participants for biomarker analyses and derivation of survival prediction model(s). Due to actual participant accrual (57) being far below the minimum required, no data were collected on the ability of models and/or biomarkers to predict time to treatment failure.
Arm/Group | R-CHOP
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Response Rate of Study Participants at the End of Protocol Therapy
Description: Rate of participants achieving complete response (CR), complete response/unconfirmed (CRu) partial response (PR) according to Non-Hodgkin's Lymphoma response criteria.
Time Frame: Up to 8 cycles, about 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | R-CHOP
Number analyzed (Participants) | 57
Participants
  Complete Response (CR) | 40
  Complete Response unconfirmed (CRu) | 0
  Partial Response (PR) | 7
  Progressive Disease (PD) | 2
  Unknown | 8

6. Secondary Outcome: Number of Participants From Whom Fixed Tissue Samples Were Collected for Future Studies.
Description: Number of participants from whom paraffin-embedded DLBCL tissue samples were collected for future studies.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- R-CHOP: Patients will receive R-CHOP for 6 to 8 cycles:
  * Rituximab 375 mg/m2 on day 1
  * Cyclophosphamide 750 mg/m2 IV on day 1
  * Doxorubicin 50 mg/m2 on day 1
  * Vincristine 1.4 mg/m2 (maximum = 2 mg) IV on day 1
  * Prednisone 100 mg orally days 1-5, repeated every 21 days.
  Rituximab: Rituximab 375 mg/m2 on day 1 for 6 to 8 cycles
  Cyclophosphamide: Cyclophosphamide 750 mg/m2 IV on day 1 for 6 to 8 cycles
  Doxorubicin: Doxorubicin 50 mg/m2 on day 1 for 6 to 8 cycles
  Prednisone: Prednisone 40 mg/m2 orally days 1-5, repeated every 21 days for 6 to 8 cycles.
  Vincristine: Vincristine 1.4 mg/m2 (maximum = 2 mg) IV on day 1 for 6 to 8 cycles
Arm/Group | R-CHOP
Number analyzed (Participants) | 57
Participants | 57

ADVERSE EVENTS:
Arm/Group | R-CHOP
All-Cause Mortality (participants affected / at risk) | 3/57
Serious Adverse Events (participants affected / at risk) | 4/57
Other Adverse Events (participants affected / at risk) | 3/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-CHOP (N=57)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Infection - Other (Infections and infestations) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-CHOP (N=57)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Cholesterol, serum-high (hypercholestremia) (Metabolism and nutrition disorders) | 1 (1) — Baseline adverse event
Constipation (Gastrointestinal disorders) | 2 (4) — Baseline adverse event
Constitutional Symptoms - Other (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) — Baseline adverse event
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) — Baseline adverse event
Headache (Nervous system disorders) | 2 (2) — Baseline adverse event
Hypertension (Vascular disorders) | 1 (1) — Baseline adverse event
Injection site reaction (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (3)
Mood alteration (Nervous system disorders) | 1 (1) — Baseline adverse event
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (2)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (diaphoresis) (General disorders) | 1 (2)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes